CLINICAL TRIAL: NCT04807621
Title: Platelets or Fibrinogen as First-line Treatment for Bleeding During Pedatric Heart Surgery: a Randomized, Controlled Trial.
Brief Title: Platelets or Fibrinogen as First-line Treatment for Bleeding During Pedatric Heart Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Fredrik Söderlund, Consultant, Anaesthesia and Intensive Care, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FS52016
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Congenital Heart Disease
Keywords: Bleeding; Coagulopathy; Heart surgery; Cardiopulmonary bypass
MeSH Terms: conditions — Heart Defects, Congenital; Hemorrhage; Hemostatic Disorders | interventions — Platelet Transfusion; Fibrinogen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelets (Active Comparator): Patients recieve, in the presence of significant bleeding and pathological results of ROTEM analysis, a platelet transfusion.
  Interventions: Biological: Platelet transfusion
- Fibrinogen (Experimental): Patients recieve, in the presence of significant bleeding and pathological results of ROTEM analysis, fibrinogen concentrate.
  Interventions: Biological: Fibrinogen concentrate

INTERVENTIONS:
Biological: Platelet transfusion — Platelets (10 ml/kg body weight) is transfused.
  Arms: Platelets
Biological: Fibrinogen concentrate — Fibrinogen concentrate (300 mg/kg body weight) is administered.
  Arms: Fibrinogen

SUMMARY:
The study aims to test whether platelet transfusion or fibrinogen concentrate is the most effective treatment of intraoperative bleeding, when performing open heart surgery with cardiopulmonary bypass on children with congenital heart defects.

ELIGIBILITY:
Inclusion Criteria:

* Children < 1 years of age, scheduled for open surgery of congenital heart defects, using cardiopulmonary bypass.
* Body weight < 10 kg.
* Expected CPB time > 90 minutes.

Exclusion Criteria:

* Known coagulation disorder, current treatment with antiplatelet and/or anticoagulant drugs, major surgery the past month before the planned surgery, preoperative kidney or liver failure (defined as creatinine and/or transaminases > normal interval for the patient´s age), gestational age < 34 weeks.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-03-14 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
HEPTEM-A10 | 45 minutes after intervention
  The outcome measure is a measure of global coagulation efficacy, obtained by ROTEM analysis.

SECONDARY OUTCOMES:
Amount of transfused packed red blood cells | up to first postoperative morning

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No